CLINICAL TRIAL: NCT06631794
Title: Evaluation of the Impact of a HPV Vaccination Talk with Third Grade Students on Their Papillomavirus Vaccination Coverage.
Brief Title: Evaluation of the Impact of a HPV Vaccination Talk with Third Grade Students
Acronym: HPV-ADO
Status: Not yet recruiting | Type: Observational
Sponsor: Hopital Foch (Other)
Collaborators: Agence Regionale de Sante d'Ile de France (Unknown); Ospharm coopérative (Unknown); French Interregional Group of Clinical Research and Innovation (Other); Communauté professionnelle territoriale de santé (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2023_0258; 2023_0258 (Other: HopitalFoch)
Record Dates: First submitted 2024-09-09; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Teenagers

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: A short talk about the importance of HPV vaccination — Investigator plan to set up a short talk to 3rd grade classes in addition to the usual sexual health training. The issue of HPV vaccination will be systematically addressed for 10 minutes to encourage catch-up vaccination.
  The usual training include different themes such us : definition of sexual health, anatomy, sexually transmitted infections contraception/condoms, menstrual cycles, voluntary interruption of pregnancy, consent, sexual abuse/violence/harassment, pornography, anti-discrimination....
  A 45-minute talk will include 2 or 3 topics from the above list. A ten minutes of talk will be added to the usual training to explain the HPV vaccination (a topic not usually addressed in sexual health training), covering the following elements: definition of HPV infection

SUMMARY:
This is a prospective pragmatic study to assess the impact of a HPV vaccination talk in secondary school on actual vaccine dispensing in test communes compared with control communes. The talk consist on a briefing on the importance of vaccination.

This is a controlled study, since two communes will benefit from the HPV vaccination talk, while the other two will serve as controls without set up of the HPV vaccination talk. The set up of this presentation will be open-label.

DETAILED DESCRIPTION:
The main aim of the present study is to investigate the impact of HPV vaccination talk with 3rd grade school children on HPV vaccine dispensing by making them actors in their own health. A significant benefit on vaccination coverage is expected. In addition, a flyer providing information and raising awareness of infections and the benefits of HPV vaccination will be sent to parents at the end of the talk.

ELIGIBILITY:
Inclusion Criteria:

* 3rd grade students enrolled in public secondary schools in Suresnes and Rueil-Malmaison.

Exclusion Criteria:

* Students absent on the day of the talk.
* Students unwilling/unable to complete questionnaire.

Ages: 14 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 3rd grade students enrolled in public secondary schools in Suresnes and Rueil-Malmaison.
Sampling Method: Probability Sample
Enrollment: 1170 (Estimated)
Dates: Start 2024-10-23 (Estimated); Primary Completion 2025-04-23 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Impact Assessement of a sexual health talk with middle school students in 3rd grade on the dispensation of HPV vaccines among young people born in 2010. | 12 months preceding the talk and the 6 months following the talk
  The aim of this study is to evaluate the impact of a sexual health talk with middle school students in 3rd grade on the dispensation of HPV vaccines among young people born in 2010.
  The main evaluation criterion for this study is the number of monthly HPV vaccine dispensations among young people born between 01/01/2010 and 31/12/2010. These data will be communicated by the OSPHARM cooperative or by pharmacies, over the 12 months preceding the talk and the 6 months following, in order to be able to assess the impact of the latter on dispensations.

SECONDARY OUTCOMES:
1rst Secondary outcoume | 8 weeks
  Evaluate the implementation of sexuality education sessions as part of middle school educational programs.
2nd Secondary outcoume | 8 weeks
  Evaluate the knowledge of Suresnes and Rueil-Malmaison 3rd grade students about HPV infection and HPV vaccination before and after the talk.
  This outcome will be evaluated through questionnaire
3rd secondary outcoume | 8 weeks
  Evaluate middle-school students; satisfaction with the HPV vaccination information talk.
  This outcome will be evaluated through questionnaire
4 th secondary outcoume | 8 weeks
  Evaluate adherence to the sexual health talk by Suresnes and Rueil-Malmaison middle schools.
  This outcome will be assessed through the mesearement of the rate of completed questionnaires
5 th secondary outcoume | 6 months after talk
  Estimating the rate of young people born in 2010 vaccinated against HPV by gender.
  The estimation rate will be calculated with data collected from the ospharm cooperative application.

IPD SHARING:
Plan to Share IPD: Undecided